CLINICAL TRIAL: NCT05815823
Title: The Effect of Virtual Reality Assisted Upper Extremity Robotic Therapy on Pain, Daily Living Activities and Functional Status in Patients With Stroke
Brief Title: Effect of Robotic Therapy on Upper Extremity With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Canan Avcı, Specialist of physical medicine and rehabilitation, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/14/01
Record Dates: First submitted 2023-03-22; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: the Effect of Virtual Reality on Stroke Rehabilitation
Keywords: stroke; upper extremity; robot-assisted therapy; armeo
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional therapy (Experimental): 20 sessions of conventional therapy was applied for 5 days a week for 4 weeks, 1 hour a day
  Interventions: Other: conventional therapy
- robot-assisted therapy (Experimental): 20 sessions of upper extremity robot-assisted therapy was applied for 4 weeks, 5 days a week, 30 minutes a day.
  Interventions: Other: robotic exercise therapy; Other: conventional therapy

INTERVENTIONS:
Other: robotic exercise therapy — Functional exercise programs such as collecting rain in a glass, grating vegetables, goalkeeper, cleaning the stove, watering flowers, wiping windows, catching fish, and exploring landscapes were applied by robotic games to the patients
  Other Names: robotic exercise
  Arms: robot-assisted therapy
Other: conventional therapy — streching, range of motion, strengthening, balance and walking exercise

SUMMARY:
The purpose of this study is to determine how adding virtual reality assisted robotic treatment to traditional rehabilitation affects stroke patients' pain levels, functional status, and daily living activities.After conventional and robotic therapy Each patient was evaluated The Barthel Index (BI), the Fugl Meyer Assessment Upper Extremity (FMA-UE), and the Visual Analogue Scale (VAS) were used to assess the patients' pain, daily living activities, and upper extremity motor function.

DETAILED DESCRIPTION:
The purpose of this study is to determine how adding virtual reality assisted robotic treatment to traditional rehabilitation affects stroke patients' pain levels, functional status, and daily living activities.

Materials and Methods: The study included 40 stroke patients. Two groups of patients were created. Group I also underwent 20 sessions of upper extremity robot-assisted therapy for 4 weeks, 5 days a week, for 30 minutes per session, in addition to receiving conventional therapy (5 days a week for 4 weeks, 1 hour each day). Group II only got traditional therapy. Each patient was assessed both before and after the procedure.

The Barthel Index (BI), the Fugl Meyer Assessment Upper Extremity (FMA-UE), and the Visual Analogue Scale (VAS) were used to assess the patients' pain, daily living activities, and upper extremity motor function.

ELIGIBILITY:
Inclusion Criteria:

- Ischemic or hemorhagic hemiplegia

* Brunnstrom upper extremity motor stage ≥3
* At least 3 months have passed
* Modified Ashworth Score ≤2
* 18-85 year old patients with diagnosis of stroke

Exclusion Criteria:

* Aphasia
* Cognitive impairment
* mini mental test <24
* deformity and / or contracture in the upper extremity
* Patients diagnosed with KBAS

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
FMA-UE scale | baseline
  FMA-UE evaluates the hemiparetic arm's mobility, including reflexes, the presence of synergies, and each of the upper limb's independent motions, including grasp. The dysmetria, coordination, and velocity of the patient are also evaluated using items on this scale. It is intended to assess muscle strength, reflex actions, and movement control in the upper extremity following a stroke. It has 33 elements and accepts values ranging from 0 to 2. Scores under 31 suggest a weak upper extremity, scores between 32 and 47 show a restricted upper extremity, scores between 48 and 52 indicate a noteworthy upper extremity, and scores between 53 and 66 indicate a full upper extremity.
FMA-UE scale | after treatment (1 month)
  FMA-UE evaluates the hemiparetic arm's mobility, including reflexes, the presence of synergies, and each of the upper limb's independent motions, including grasp. The dysmetria, coordination, and velocity of the patient are also evaluated using items on this scale. It is intended to assess muscle strength, reflex actions, and movement control in the upper extremity following a stroke. It has 33 elements and accepts values ranging from 0 to 2. Scores under 31 suggest a weak upper extremity, scores between 32 and 47 show a restricted upper extremity, scores between 48 and 52 indicate a noteworthy upper extremity, and scores between 53 and 66 indicate a full upper extremity.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP